CLINICAL TRIAL: NCT01498354
Title: Comparing the Efficiency of Two Dimensional High Definition (TEO) Versus Three Dimensional (TEM) Endoscopic Systems in Transanal Endoscopic Surgery; a Prospective Control Trial
Brief Title: Efficiency of Two Dimensional High Definition vs Three Dimensional Endoscopic Systems in Transanal Endoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Medical Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEO-TEM-2010-01
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Rectal Adenoma
Keywords: Transanal endoscopic microsurgery; Transanal endoscopic operations; Rectal adenomas; Transanal endoscopic surgery; Rectal adenocarcinomas "in situ"
MeSH Terms: interventions — Transanal Endoscopic Microsurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2-D high definition TEO (transanal endoscopic operation) (Experimental)
  Interventions: Procedure: 2-D high definition vision systems, transanal endoscopic operation (TEO)
- Transanal endoscopic microsurgery (TEM) (Active Comparator): Transanal endoscopic microsurgery (TEM), 3-D vision system using a rectoscope, which allows access to rectal tumors located up to 20 cm from the anal verge
  Interventions: Procedure: Transanal endoscopic microsurgery (TEM)

INTERVENTIONS:
Procedure: 2-D high definition vision systems, transanal endoscopic operation (TEO) — Transanal endoscopic operation (TEO). Through its 2-D vision system using a rectoscope, this procedure allows access to rectal tumors located up to 20 cm from the anal verge
  Arms: 2-D high definition TEO (transanal endoscopic operation)
Procedure: Transanal endoscopic microsurgery (TEM) — Transanal endoscopic microsurgery (TEM). 3-D vision system using a rectoscope, allowing access to rectal tumors located up to 20 cm from the anal verge
  Arms: Transanal endoscopic microsurgery (TEM)

SUMMARY:
Introduction: The usual surgical technique for large adenomatous tumors and rectal cancer is anterior resection of the rectum or abdominoperineal resection. These techniques are associated with high mortality and morbidity and with genitourinary dysfunctions.

To solve these problems, transanal endoscopic microsurgery (TEM) was designed. Through its 3-D vision system using a rectoscope, this procedure allows access to rectal tumors located up to 20 cm from the anal verge. It is associated with minimal morbidity and has few repercussions for anal continence.

The use of 2-D high definition cameras and screens obtains images of a similar quality to 3-D images. This means that from the surgical point of view the procedure known as TEO (transanal endoscopic operation) seems as practicable as classic TEM.

Main aim: To assess the effectiveness of 2-D high definition vision systems (TEO) versus conventional 3-D (TEM) in endoscopic surgery of rectal tumors, with respect to surgical facility, postoperative morbidity, quality of the surgical specimens, and cost.

Design: Prospective, controlled, randomized study of the efficacy of the use of 2-D high definition endoscopic systems versus 3-D (TEM) in transanal endoscopic surgery.

Disease studied: Rectal adenomas and adenocarcinomas "in situ" suitable for local surgery.

Main variable evaluated: Cost per procedure assuming similar surgical efficacy and equal postoperative morbidity.

Study population and total number of patients: Patients diagnosed with rectal tumor treated with curative intent (rectal adenomas and adenocarcinomas "in situ"). The total sample calculated for the trial was 36 patients, 18 in each group (TEO and TEM).

Timing and expected finish date: After approval by the CEIC, the expected date for the inclusion of the first patient was August 2010. The study is expected to last 18-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex older than 18 years
* Rectal tumor identified as rectal adenoma by multifocal biopsy using colonoscopy, with endorectal ultrasound and magnetic resonance imaging findings of non-invasive tumor.
* Size of the tumor between 2 and 6 cm in maximum diameter.
* Tumor location, lower edge at least 2 cm from the anal verge, and upper edge at least 15 cm from the anal verge.
* ASA score more than III.
* intervention was performed under general anesthesia

Exclusion Criteria:

* Invasive adenocarcinoma shown in the final pathology study. "in situ" or intraepithelial adenocarcinomas are not excluded .
* Pregnant patients
* Patients with liver cirrhosis or blood dyscrasia.
* Patients who can not be administered under general anesthesia.
* Patients on antiplatelet or anticoagulation therapy who have not been properly prepared for surgery.
* Presence of two or more transanal endoscopic excisions in the same procedure.
* Informed consent not signed.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Cost per procedure assuming similar surgical efficacy and equal postoperative morbidity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Serra-Aracil, MD, Principal Investigator — Corporacion Sanitaria Universitaria Parc Tauli
Locations (1):
- Corporacion Sanitaria Universitaria Parc Tauli, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Serra-Aracil X, Mora-Lopez L, Alcantara-Moral M, Caro-Tarrago A, Navarro-Soto S. Transanal endoscopic microsurgery with 3-D (TEM) or high-definition 2-D transanal endoscopic operation (TEO) for rectal tumors. A prospective, randomized clinical trial. Int J Colorectal Dis. 2014 May;29(5):605-10. doi: 10.1007/s00384-014-1849-3. Epub 2014 Mar 28. PMID 24676506